CLINICAL TRIAL: NCT06367699
Title: Conversational Agents to Improve HPV Vaccine Acceptance in Primary Care
Brief Title: Conversational Agents to Improve HPV Vaccine Acceptance in Primary Care (ECA-HPV)- Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were informed by the NCI that this research no longer aligns with NCI values, therefore our grant was terminated and we had received a stop work order.
Sponsor: Tufts Medical Center (Other)
Collaborators: Boston Medical Center (Other); Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-44821
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Human Papilloma Virus
Keywords: Human Papilloma Virus; Cancer Prevention; Vaccination Promotion; Vaccination Attitudes; Vaccination Completion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Usual Care (Active Comparator): An internet-based measure, REDCap, will be used for parent/guardian and adolescent participants to complete surveys at baseline, after the index well child visit, and after the second well child visit. Both parent/guardian and adolescent participants do not have access to the ECA-HPV app. Adolescent participants will receive usual standard of care.
  Interventions: Behavioral: Usual Care
- ECA-HPV App with Clinic Notification and Adolescent Functions Disabled (Experimental): The ECA-HPV (Embodied Conversational Agent adapted for this project) system comprises of a smartphone-based ECA parent/guardian interface, where the parent/guardian participants can receive HPV vaccine promotion and counseling from an interactive agent. The clinic notification feature is disabled on the app. Adolescent participants do not receive the adolescent version of the ECA-HPV app. An internet-based measure, REDCap, will be used for parent/guardian and adolescent participants to complete surveys at baseline, after the index well child visit, and after the second well child visit.
  Interventions: Behavioral: ECA-HPV App with Clinic Notification and Adolescent Functions Disabled
- ECA-HPV App with Clinic Notification Function Enabled (Experimental): The ECA-HPV (Embodied Conversational Agent adapted for this project) system comprises of a smartphone-based ECA parent/guardian interface, where the parent/guardian participants can receive HPV vaccine promotion and counseling from an interactive agent. With the clinic notification function enabled, parent/guardian participants can communicate their concerns, questions, and logistical barriers to the clinic staff. Adolescent participants do not receive the adolescent version of the ECA-HPV app. An internet-based measure, REDCap, will be used for parent/guardian and adolescent participants to complete surveys at baseline, after the index well child visit, and after the second well child visit.
  Interventions: Behavioral: ECA-HPV App with Clinic Notification Function Enabled
- ECA-HPV App with Adolescent Function Enabled (Experimental): The ECA-HPV (Embodied Conversational Agent adapted for this project) system comprises of a smartphone-based ECA parent/guardian interface, where the parent/guardian participants can receive HPV vaccine promotion and counseling from an interactive agent. Adolescent participants receive the adolescent version of the ECA-HPV app, which includes age-appropriate education and adolescent-focused engagement features, like games. The clinic notification feature is disabled on both the parent/guardian and adolescent apps. An internet-based measure, REDCap, will be used for parent/guardian and adolescent participants to complete surveys at baseline, after the index well child visit, and after the second well child visit.
  Interventions: Behavioral: ECA-HPV App with Adolescent Function Enabled
- ECA-HPV App with Clinic Notification and Adolescent Functions Enabled (Experimental): Participants will receive the full ECA-HPV (Embodied Conversational Agent adapted for this project) system on their smartphone app, which includes both the clinic notification and adolescent functions enabled. With the clinic notification function enabled, parent/guardian participants can communicate their concerns, questions, and logistical barriers to the clinic staff. Adolescent participants receive the adolescent version of the ECA-HPV app, which includes age-appropriate education and adolescent-focused engagement features, like games. An internet-based measure, REDCap, will be used for parent/guardian and adolescent participants to complete surveys at baseline, after the index well child visit, and after the second well child visit.
  Interventions: Behavioral: ECA-HPV App with Clinic Notification and Adolescent Functions Enabled

INTERVENTIONS:
Behavioral: Usual Care — Parent/guardian and adolescent participants will not receive the ECA-HPV system intervention. A survey will be given via REDCap to the parent/guardian and adolescent participants at baseline, after the first well child clinic visit, and after the second well child clinic visit to assess self-reported vaccination attitudes and behaviors. Adolescent participants will receive usual care.
  Arms: Usual Care
Behavioral: ECA-HPV App with Clinic Notification and Adolescent Functions Disabled — Parent/guardian participants will interact with the ECA-HPV smartphone-based system over a period of ~16 months. The ECA-HPV is designed to interact with parents/guardians to increase vaccine acceptability prior to the clinic visit. A survey will be given via REDCap at baseline, after the first well child clinic visit, and after the second well child clinic visit to both the parent/guardian and adolescent to assess self-reported vaccination attitudes and behaviors. Parent/guardian participants will also be asked questions about the ECA-HPV app. The clinic notification and adolescent functions of the complete ECA-HPV app are disabled. Adolescent participants will receive usual care.
  Arms: ECA-HPV App with Clinic Notification and Adolescent Functions Disabled
Behavioral: ECA-HPV App with Clinic Notification Function Enabled — Parent/guardian participants will interact with the ECA-HPV smartphone-based system over a period of ~16 months. The ECA-HPV is designed to interact with parents/guardians to increase vaccine acceptability prior to the clinic visit. A survey will be given via REDCap at baseline, after the first well child clinic visit, and after the second well child clinic visit to both the parent/guardian and adolescent to assess self-reported vaccination attitudes and behaviors. Parent/guardian participants will also be asked questions about the ECA-HPV app and the clinic notification feature. The clinic notification is enabled on the parent/guardian ECA-HPV app, however, the adolescent does not have access to the adolescent ECA-HPV app. Adolescent participants will receive usual care.
  Arms: ECA-HPV App with Clinic Notification Function Enabled
Behavioral: ECA-HPV App with Adolescent Function Enabled — Parent/guardian participants will interact with the ECA-HPV smartphone-based system over a period of ~16 months. The ECA-HPV is designed to interact with parents/guardians to increase vaccine acceptability prior to the clinic visit. A survey will be given via REDCap at baseline, after the first well child clinic visit, and after the second well child clinic visit to both the parent/guardian and adolescent to assess self-reported vaccination attitudes and behaviors as well as ECA-HPV app use and satisfaction. The adolescent function is enabled, however, the clinic notification function is disabled. Thus, the ECA-HPV system app will have an adolescent-facing feature for adolescent participants to engage with the agent. Adolescent participants will receive usual care and will be able to engage with the adolescent version of the ECA-HPV app throughout the duration of the study.
  Arms: ECA-HPV App with Adolescent Function Enabled
Behavioral: ECA-HPV App with Clinic Notification and Adolescent Functions Enabled — Parent/guardian participants will interact with the complete ECA-HPV smartphone-based system over a period of ~16 months. The ECA-HPV is designed to interact with parents/guardians to increase vaccine acceptability prior to the clinic visit. A survey will be given to parent/guardian participants via REDCap at baseline, after the first well child clinic visit, and after the second well child clinic visit to both the parent/ guardian and adolescent to assess self-reported vaccination attitudes and behaviors as well as ECA-HPV app use and satisfaction and questions about the clinic notification feature. The complete ECA-HPV app includes the parent version and adolescent versions of the ECA-HPV app. Both versions have the clinic notification feature enabled. Adolescent participants will receive usual care and can engage with the adolescent version of the ECA-HPV app throughout the study.
  Arms: ECA-HPV App with Clinic Notification and Adolescent Functions Enabled

SUMMARY:
The objective of this study is to assess the use of and satisfaction with the ECA-HPV intervention over a 16-month period, its ability to increase HPV vaccination, and the comparative effectiveness of clinic notification and adolescent ECA components on these factors.

DETAILED DESCRIPTION:
In the US, universal Human Papillomavirus (HPV) vaccination has the potential to decrease overall burdens of certain cancers. However, HPV vaccination rates for US adolescents of all races, ethnicities, and income levels remain below national targets. Embodied Conversational Agents (ECAs) are animated computer agents that simulate face-to-face conversation between a patient and a caregiver, to provide a natural and intuitive computer interface that is accessible to patients of all levels of health and computer literacy. In this project, we produced smartphone ECAs for HPV vaccination to provide vaccine recommendations and motivational interviewing to parents/guardians and vaccine-eligible adolescents and facilitate communication with clinic staff.

In this study, we will be using the ECA-HPV system to administer interactive information to parents and adolescents in the form of a smartphone app. We will obtain data from participants by asking subjects to fill out surveys on REDCap and electronically from use of the ECA system. The parent/guardian and adolescent participants will each complete 3 surveys over a 16-month period occurring at baseline, after the first well child visit, and after the second well child visit (anticipated to be ~1 year after their initial well child visit). Additionally, a randomly selected subset of adolescent and parent/guardian participant dyads who were in an intervention group where adolescents also had the ECA-HPV adolescent app will be interviewed after their first well child visit about their experience. Lastly, for healthcare providers who have interacted with at least 5 study participants in any of the intervention groups, they will be recruited to participate in qualitative interviews.

For this RCT, the participant dyads (parent/guardian and adolescent) will be randomly assigned into one of five groups (N = 875 dyads). The control group will receive usual standard care (n = 175 dyads). The other four groups are intervention groups in which all will get the ECA-HPV app for the parent/guardian. Additionally, these four groups will receive either (1) the complete ECA-HPV, including the ECA-HPV adolescent app and the clinic notification feature (on both the parent/guardian and adolescent apps) (n = 175 dyads), (2) the ECA-HPV app and adolescent ECA-HPV app with the clinic communication function disabled (n = 175 dyads), (3) the ECA-HPV app with clinic notification with no adolescent ECA-HPV app (n = 175 dyads), or (4) the ECA-HPV app with no clinic communication feature and no adolescent ECA-HPV app (n = 175 dyads).

For this study, we will evaluate whether (1) adolescents who receive the ECA-HPV intervention will have a higher rate of HPV vaccine series completion, (2) participating parents/guardians will have higher vaccine knowledge and greater intention to vaccinate, and (3) vaccine series completion rates will be higher for those receiving the full ECA-HPV intervention, compared to those who get ECA-HPV without the adolescent or clinic notification components.

ELIGIBILITY:
Inclusion Criteria:

For parent/guardian participants:

1. Speaks English fluently
2. Able to independently consent
3. Has adequate corrected vision to use the ECA-HPV system (based on their ability to go through the consent form)
4. Has adequate hearing to use the ECA-HPV system (based on their ability to hear the research staff member conducting the consent process)
5. Has a smartphone that is able to support the ECA-HPV app

For adolescent participants:

1. Is between the ages of 9-12 at the time of the index (first) well child visit
2. Has received either 1 or none of the HPV vaccine series
3. Speaks English fluently
4. Able to independently assent
5. Has adequate corrected vision to use the ECA-HPV system
6. Has adequate hearing to use the ECA-HPV system
7. Has a smartphone or has access to parent/guardian's smartphone (that is able to support the ECA-HPV app)
8. Has an upcoming well child visit at Boston Medical Center

Exclusion Criteria (for all participants):

1. Is not able to use the ECA-HPV system
2. Has already participated in the study before

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
HPV vaccination series completion comparing the control group to the intervention groups | 16 months
  HPV vaccination series completion for the control group will be compared to the collective rate for the intervention groups. A review of medical records at the T2 timepoint will be done for vaccination series completion.
HPV vaccination series completion comparing the intervention groups | 16 months
  HPV vaccination series completion will be assessed between participants randomized to the full ECA-HPV versus people randomized to the ECA-HPV with no adolescent app function and no clinic notification function. A review of medical records at the T2 timepoint will be done for vaccination series completion.

SECONDARY OUTCOMES:
HPV Knowledge | 16 months
  The parent/guardian participants will be asked questions about their HPV knowledge in all three surveys: at baseline (T0), post-first well child visit (T1), and post-second well child visit (T2). Participants will fill out the surveys in REDCap. The outcomes for this measure at T1 and T2 will be compared to the outcome at T0.
HPV Attitudes | 16 months
  Both the parent/guardian and adolescent participants will be asked questions about their attitudes towards HPV in all three surveys: at baseline (T0), post-first well child visit (T1), and post-second well child visit (T2). Participants will fill out these surveys in REDCap. The outcomes for this measure at T1 and T2 will be compared to the outcome at T0.
General Vaccine Attitudes | 16 months
  The parent/guardian participants will be asked questions about their attitudes towards vaccines in general in all three surveys: at baseline (T0), post-first well child visit (T1), and post-second well child visit (T2). Participants will fill out these surveys in REDCap. The outcomes for this measure at T1 and T2 will be compared to the outcome at T0.
ECA-HPV App Satisfaction | 16 months
  If participants are in an intervention group with the ECA-HPV app, their post-first well child visit survey will include questions about use and satisfaction of the app. Participants will fill out these surveys in REDCap.
Clinic Notification Feature Satisfaction | 16 months
  If participants are in an intervention group with the ECA-HPV app and the clinic notification function enabled, their post-first well child visit survey will include questions about use and satisfaction of this feature. Participants will fill out these surveys in REDCap

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No